CLINICAL TRIAL: NCT04494997
Title: Dentists' Perception Regarding the Use of Social Media for Professional Purpose: A Cross-sectional Study
Brief Title: Dentists' Perception Regarding the Use of Social Media for Professional Purpose
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Dr Shiva Shankar Bugude, Assistant Professor, Qassim University
Other Study IDs: QassimU1
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Social Media; Perception, Self
Keywords: Social Media; Dentists; Perception; Professional purpose
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dentists: Practicing Dental Health Professionals who are either General Dentists &/or Specialists Dentists are part of the Cohort. They should have held or currently hold Social Media account for their Professional purpose. They should have used or currently using their Social Media account for Professional purpose. The Google form questionnaire survey link will be shared with the Dentists in internet via Social Media &/Or email to seek responses. The link will be available for single response for a single respondent.
  Interventions: Other: Survey Questionnaire

INTERVENTIONS:
Other: Survey Questionnaire — This Cross sectional study uses Questionnaire with Closed ended questions. The survey form is designed using Google forms program. Survey initial question seeks CONSENT from the respondent. Survey collects data under 4 sections.
  Section I: Demographic details Section II: 6 Questions regarding use of your Social Media for Professional activities.
  Section III: 7 Questions regarding the advantages of your Social Media use. Section IV: 5 Questions regarding the disadvantages of your Social Media use.
  The Google form questionnaire survey link will be shared with the Dentists in internet via Social Media &/Or email to seek responses. The link will be available for single response for a single respondent.

SUMMARY:
Social Media has significant influence in everyone's life. Social media is considered as one of the biggest revolution in the information technology. It empowers the users to express and share their thoughts, opinions, views, and content to the rest of the world. Entire world id just a click away from the Social Media users. Social media gives an immense opportunity to grow through right connectivity and collaboration. Healthcare professionals are no exception for this. Healthcare professionals can make appropriate use of Social media for public outreach with their content and educate them. Social Media with its tools enables the professionals to create multimedia content to engage the audiences. It also improves professional connectivity and better public display of professional skills. These can enhance the professional growth through public availability and accessibility. Social Media giants in the recent times were also blamed for data privacy and protection. There are issues of excessive indulgence into privacy through access of users' locations and contacts. Overt advertisements and unnecessary tagging to the content by unknown users cannot be ignored. Our cross sectional study is aimed to understand Dentist' perspective at professional level, regarding their use, advantages and disadvantages of Social Media.

DETAILED DESCRIPTION:
Objectives of the Study:

To understand which Social Media platform is used the most by the Dentists for their Professional purpose.

To understand the different uses of Social Media by the Dentists for their Professional purpose.

To understand the Dentists' perspective of the ADVANTAGES of their SOCIAL MEDIA accounts for their Professional purpose.

To understand the Dentists' perspective of the DISADVANTAGES of their SOCIAL MEDIA accounts for their Professional purpose.

Sample Size Sample size calculated using OpenEpi, Version 3, open source calculator. n-384, Confidence Interval 95%, Design Effect -1, anticipated % frequency - 50%.

Methodology This Cross sectional study uses Questionnaire with Closed ended questions. The survey form is designed using Google forms program. Survey initial question seeks CONSENT from the respondent. Survey collects data under 4 sections.

Section I: Demographic details Section II: 6 Questions regarding use of your Social Media for Professional activities.

Section III: 7 Questions regarding the advantages of your Social Media use. Section IV: 5 Questions regarding the disadvantages of your Social Media use.

Section III & IV involves exclusive use of Likert Scale questions.

ELIGIBILITY:
Inclusion Criteria:

Dentists who currently hold Social Media account/accounts & use for Professional activity.

Dentists who held Social Media account/accounts & used for Professional activity.

Dentists who create their OWN MULTIMEDIA NEW CONTENT in Social Media. Dentists who share &/Post Profession related text posts in Social Media. Dentists who share &/Post Profession related pictures in Social Media. Dentists who share &/Post Profession related videos in Social Media.

Exclusion Criteria:

Dentists who never held social media account. Dentists who use social media exclusive for Personal purpose. Dentists who never used social media for Professional purpose.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Practicing Dental Health Professionals who are either General Dentists &/or Specialists Dentists are part of the Cohort. They should have held or currently hold Social Media account for their Professional purpose. They should have used or currently using their Social Media account for Professional purpose. The Google form questionnaire survey link will be shared with the Dentists in internet via Social Media &/Or email to seek responses. The link will be available for single response for a single respondent.
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Perception of Social Media advantages | 15th of August 2020
  The primary outcome of the Dentists perception regarding the advantages of their Social Media account use for Professional purpose would be analysed by data interpretation obtained from Section III of the survey responses.
Perception of Social Media disadvantages | 15th of August 2020
  The primary outcome of the Dentists perception regarding the disadvantages of their Social Media account use for Professional purpose would be analysed by data interpretation obtained from Section IV of the survey responses.
Perception of Social Media use | 15th of August 2020
  The primary outcome of the Dentists perception regarding the advantages of their Social Media account use for Professional purpose would be analysed by data interpretation obtained from Section II of the survey responses.

SECONDARY OUTCOMES:
Correlation of type of practice & Social media use | 15th of August 2020
  Correlation of the Dentists' type of practice data (Rural/Urban) will be correlated with the data of the use of Social Media use. Necessary statistical tests will be used to find out the significance level at p-value 0.05.
Correlation of Age & Social media use | 15th of August 2020
  Correlation of the Dentists' Age data will be correlated with the data of the use of Social Media use. Necessary statistical tests will be used to find out the significance level at p-value 0.05.
Correlation of Professional qualification & Social media use | 15th of August 2020
  Correlation of the Dentists' Professional qualification data (General dentist/Specialist dentist) will be correlated with the data of the use of Social Media use. Necessary statistical tests will be used to find out the significance level at p-value 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr B Shiva Shankar, Ar Rass, Al Qassim, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The Research data will be available to the Principal Investigator. On requirement the data will be shared to whomsoever after consultation with the concerned higher authorities in the College of Applied Health sciences in Ar rass. The descriptive & analytical data will be used for scientific publication.